CLINICAL TRIAL: NCT03417960
Title: An Open Label Study to Assess the Feasibility and Tolerability of Accelerated Theta Burst Repetitive Transcranial Magnetic Stimulation (iTBS-rTMS) for the Treatment of Post-Partum Depression
Brief Title: Accelerated iTBS for Post Partum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kevin Caulfield, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00073886
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-03

CONDITIONS: Post Partum Depression
Keywords: post partum depression; theta burst; transcranial magnetic stimulation
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Open label pilot
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- iTBS (Experimental): accelerated iTBS to Left DLPFC
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — The investigators will treat post-partum depressed subjects with accelerated intermittent theta burst stimulation. iTBS will be delivered via a MagVenture MagPro100 and Cool-B65 coil. The investigators will use a standard resting motor threshold (rMT) determination to determine the TMS dose. Treatment will be delivered at 120% of the motor threshold.
  In study 1, the accelerated paradigm will consist of 10 such sessions separated by 15 minutes, for three treatment days per week. There will be 2 weeks of 10 sessions on each of three days for a total of six treatment days, divided by one treatment-free week between treatment weeks. In study 2, the accelerated paradigm will consist of 12 sessions per day for 5 total treatment days. Treatments will be delivered at the 10-20 EEG coordinate for F3 (approximating the left DLPFC), and will be found using the Beam-F3 method.

SUMMARY:
Study 1: The investigators are studying the feasibility and tolerability of 10x/day intermittent theta burst (excitatory) transcranial magnetic stimulation to the left dorsolateral prefrontal cortex over the course of 6 days for women with post-partum depression. The investigators further aim to characterize the anticipated anti-depressant effect of this treatment paradigm.

Study 2: The investigators are studying the feasibility and tolerability of 12 sessions/day of intermittent theta burse (excitatory) transcranial magnetic stimulation to the left dorsolateral prefrontal cortex over 5 days for women with post-partum depression. The investigators aim to compare the two different treatment schedules.

DETAILED DESCRIPTION:
Study 1: This is an open-label study designed to investigate the feasibility and tolerability of a novel TMS treatment protocol to treat depression in women with post-partum depression. It is known that TMS can effectively treat depression. The FDA approved protocol lasts 6 weeks and is not feasible for many women with post-partum depression. The investigators are investigating a 6 day treatment for depression which may be more acceptable for this population. The investigators further aim to characterize the ant-depressant effect of this protocol in order to design a larger trial.

Study 2: In part 2 of this study, the treatment schedule is 12 sessions over 5 days that can be completed with 8. All other procedures, inclusion/exclusion criteria, and number of total pulses delivered is the same as study 1.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Participants must be over the age of 18.
3. Participants must meet criteria for post-partum depression: a) onset of symptoms in the first year postpartum
4. Participants must have a HRSD17 greater than or equal to 14 at baseline.

Exclusion Criteria:

1. Participants must not be pregnant.
2. Participants must not meet moderate or severe use disorder of any substance with the exception of Tobacco Use Disorder.
3. Participants must not have current psychotic symptoms.
4. Participants must not have a history of dementia or other cognitive impairment.
5. Participants must not have active suicidal ideation requiring hospitalization or a suicide attempt within the past 3 months.
6. Participants must not have any contraindications to receiving rTMS (e.g. metal implanted above the neck, history of seizure, any known brain lesion).
7. Participants must not have any unstable general medical conditions.
8. Participants must not have had eclampsia during pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility and tolerability of accelerated iTBS for postpartum depression. The investigators hope to retain >80% of recruited patients (feasibility) and reach a full treatment dose of 120%rMT in >80% of enrolled women (tolerability). | 7 days
  Determine feasibility and tolerability of accelerated iTBS for postpartum depression. The investigators hope to retain >80% of recruited patients (feasibility) and reach a full treatment dose of 120%rMT in >80% of enrolled women (tolerability).

SECONDARY OUTCOMES:
Anti-depressant effect | 4 weeks
  Determine the preliminary anti-depressant effect size of a course of accelerated iTBS for women with postpartum depression. We hypothesize that at least 30% of post-partum depressed subjects receiving accelerated iTBS will achieve a response (50% reduction in symptoms as measured on Ham-D) at 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No